CLINICAL TRIAL: NCT00616187
Title: Oral High-Dose Atorvastatin Treatment in Relapsing-Remitting Multiple Sclerosis
Brief Title: Atorvastatin in Relapsing-Remitting Multiple Sclerosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: German Research Foundation (Other); German Federal Ministry of Education and Research (Other Government); Pfizer (Industry)
Responsible Party: Professor Frauke Zipp, Cecilie Vogt Clinic for Neurology, Charite University, Berlin, Germany
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1931/Si.270 am 8.5.03; ATV-D-03-007G
Record Dates: First submitted 2008-02-05; First posted 2008-02-15 (Estimated); Last update posted 2018-03-20 (Actual); Status verified 2017-12

CONDITIONS: Relapsing Remitting Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- interferon (Active Comparator)
  Interventions: Drug: interferon beta treatment to add-on atorvastatin treatment
- untreated (Sham Comparator)
  Interventions: Drug: untreated to atorvastatin treatment

INTERVENTIONS:
Drug: interferon beta treatment to add-on atorvastatin treatment — IFN-β-1a 22 µg s.c. 3 times weekly or IFN-β-1b s.c. every other day (3 months baseline) and add on oral daily 80 mg atorvastatin (9 months add on treatment)
  Arms: interferon
Drug: untreated to atorvastatin treatment — no treatment(3 months baseline)and oral daily 80 mg atorvastatin (9 months add on treatment)
  Arms: untreated

SUMMARY:
A phase II open-label baseline-to-treatment trial was designed to evaluate the safety, tolerability and efficacy of orally administered atorvastatin in patients with relapsing-remitting multiple sclerosis (RRMS). Patients with at least one gadolinium-enhancing lesion (CEL) at screening by magnetic resonance imaging (MRI) were eligible for the study. Patients are screened and enrolled in the outpatient clinic of the Cecilie Vogt Clinic at the Charité - University Medicine Berlin. After a baseline period of 3 monthly MRI scans (months -2 to 0), patients followed a 9-month treatment period on 80 mg atorvastatin daily. The primary endpoint is the number of CEL in treatment months 6 to 9 compared to baseline. Secondary endpoints include other MRI-based parameters and changes in clinical scores and immune responses.

ELIGIBILITY:
Inclusion Criteria:

* 18 - 55 years old
* MS diagnosis according McDonald criteria
* Relapsing-remitting MS
* EDSS 0 - 6
* Disease activity as occurrence of CEL in brain MRI
* IFN-beta therapy for at least 6 months

Exclusion Criteria:

* Primary chronic progressive MS
* Symptoms and signs of clinical disease conditions similar to MS
* Conditions that can disturb MRI measurements
* Clinically relevant GI diseases eg Colitis ulcerosa, Crohns disease, history of Ulcus pepticum
* Clinically relevant lung, heart, CNS, infectious disease
* Clinically relevant liver, kidney or bone marrow abnormalities (as defined by specific clinical chemistry values)
* Allergies towards Gd-DTPA
* Allergies towards constituents of the therapeutic agent
* Recruitment to other clinical trials within 6 months prior to or during this study
* Pretreatment with complete lymph irradiation, antibody therapy against lymphocyte populations (eg. anti-CD4, Campath-1H), mitoxantrone, cyclophosphamide, cyclosporin A, human antibodies, all immunomodulatory or immunosuppressive agents including recombinant cytokines or other potential experimental MS therapies (6 months prior to study start), glatiramer acetate, azathioprine, IVIg (6 months prior to study start) pregnancy or lactation
* Alcohol or drug abuse
* Inhibitors of Cytochrom P 450 3A (eg. cyclosporin, macrolide antibiotics, azole antimycotics).
* Medical or psychological conditions that could hamper with the patients capacity to understand patient information, to give the informed consent, to adhere to the protocol of the study and to be able to complete the study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2003-10; Primary Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
number of MRI contrast enhancing lesions | treatment months 6 to 9 compared to baseline

SECONDARY OUTCOMES:
other MRI-based parameters (CEL volume, T2-lesion load, T1-hypointense lesion volume, whole brain magnetization transfer ratio, and apparent diffusion coefficient of normal appearing white matter) | treatment months 6 to 9 compared to baseline

CONTACTS AND LOCATIONS:
Overall Officials: Frauke Zipp, MD, Principal Investigator — Cecilie Vogt Clinic for Neurology, Charite, Berlin

REFERENCES:
- [Derived] Paul F, Waiczies S, Wuerfel J, Bellmann-Strobl J, Dorr J, Waiczies H, Haertle M, Wernecke KD, Volk HD, Aktas O, Zipp F. Oral high-dose atorvastatin treatment in relapsing-remitting multiple sclerosis. PLoS One. 2008 Apr 9;3(4):e1928. doi: 10.1371/journal.pone.0001928. PMID 18398457